CLINICAL TRIAL: NCT03361566
Title: Einfluss Des Energy Flux Auf Die Kurzfristige Regulation Der Energie- Und Makronährstoffbilanz
Brief Title: Short-term Regulation of Energy and Macronutrient Balance: Impact of Energy Flux
Acronym: EF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: EF2016
Record Dates: First submitted 2017-10-09; First posted 2017-12-05 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Healthy
Keywords: physical activity; energy balance; caloric restriction; overfeeding; appetite regulation
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Energy Intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- low energy flux at ad libitum energy intake (Experimental): physical activity: inactive energy intake: ad libitum
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- medium energy flux at ad libitum energy intake (Experimental): physical activity: medium (3 x 55 min treadmill running at 4 km/h) energy intake: ad libitum
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- high energy flux at ad libitum energy intake (Experimental): physical activity: high (3 x 110 min treadmill running at 4 km/h) energy intake: ad libitum
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- Low energy flux at energy balance (Experimental): physical activity: inactive energy intake: individual energy balance
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- medium energy flux at energy balance (Experimental): physical activity: medium (3 x 55 min treadmill running at 4 km/h) energy intake: individual energy balance
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- high energy flux at energy balance (Experimental): physical activity: high (3 x 110 min treadmill running at 4 km/h) energy intake: individual energy balance
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- low energy flux at caloric restriction (Experimental): physical activity: inactive energy intake: caloric restriction -25%
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- medium energy flux at caloric restriction (Experimental): physical activity: medium (3 x 55 min treadmill running at 4 km/h) energy intake: caloric restriction -25%
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- high energy flux at caloric restriction (Experimental): physical activity: high (3 x 110 min treadmill running at 4 km/h) energy intake: caloric restriction -25%
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- low energy flux at overfeeding (Experimental): physical activity: inactive energy intake: overfeeding +25%
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- medium energy flux at overfeeding (Experimental): physical activity: medium (3 x 55 min treadmill running at 4 km/h) energy intake: overfeeding +25%
  Interventions: Behavioral: physical activity; Behavioral: energy intake
- high energy flux at overfeeding (Experimental): physical activity: high (3 x 110 min treadmill running at 4 km/h) energy intake: overfeeding +25%
  Interventions: Behavioral: physical activity; Behavioral: energy intake

INTERVENTIONS:
Behavioral: physical activity — 3 different levels of physical activity
Behavioral: energy intake — 4 different types of energy intake

SUMMARY:
Aim of the study is to investigate the impact of energy flux (achieved by changes in physical activity) under the conditions of energy balance, caloric restriction and overfeeding in healthy subjects.

DETAILED DESCRIPTION:
A low energy flux is achieved by low energy expenditure, equivalent to low physical activity and with a corresponding low energy intake. A high energy flux is achieved by high energy expenditure, equivalent to high physical activity and with a corresponding high energy intake, respectively.

The protocol of this randomized, intra-individual nutrition intervention includes 12 one-day interventions with 3 different levels of energy flux and 4 different diet conditions.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years of age
* healthy
* BMI between 18.5 and 31 kg/m2

Exclusion Criteria:

* smoking
* food allergies
* alternative nutrition habits like vegetarian / vegan
* chronic diseases
* regular medication intake
* claustrophobia
* weight loss > 5 kg in the last 3 years

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
energy balance | 24 hours
  difference between predefined energy balance and measured energy balance

SECONDARY OUTCOMES:
ghrelin levels | every 2 hours during the day over 14 hours
  area under the curve of total plasma ghrelin
arterial stiffness | 15 hours
  pulse wave velocity

CONTACTS AND LOCATIONS:
Overall Officials: Anja Bosy-Westphal, Prof PhD MD, Principal Investigator — University of Hohenheim, Stuttgart, Germany
Locations (1):
- Institute of Nutritional Medicine, University of Hohenheim, Stuttgart, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hagele FA, Busing F, Nas A, Hasler M, Muller MJ, Blundell JE, Bosy-Westphal A. Appetite Control Is Improved by Acute Increases in Energy Turnover at Different Levels of Energy Balance. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4481-4491. doi: 10.1210/jc.2019-01164. PMID 31305927